CLINICAL TRIAL: NCT06916780
Title: Elhafez Technique Combined With Dynamic Scapulohumeral Mobilization in Patients With Shoulder Adhesive Capsulitis
Brief Title: Elhafez Technique Combined With Dynamic Scapulohumeral Mobilization in Shoulder Adhesive Capsulitis
Acronym: DSM
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: For a public vacation
Sponsor: Haytham M Elhafez (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Haytham M Elhafez, Professor of Physical Therapy, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/004/007724
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Adhesive Capsulitis of the Shoulder
Keywords: Elhafez technique; Adhesive capsulitis; Dynamic scapulohumeral mobilization
MeSH Terms: conditions — Bursitis | interventions — Lasers; High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Active Comparator): Participants will receive traditional physical therapy (ultrasonic, laser, exercises and home program)
  Interventions: Other: Laser and ultrasound
- Elhafez Technique Group (Experimental): Participants will receive Elhafez technique only
  Interventions: Other: Laser and ultrasound
- Elhafez Technique and DSM Group (Experimental): Participants will receive Elhafez technique and dynamic scapulohumeral mobilization
  Interventions: Other: Laser and ultrasound

INTERVENTIONS:
Other: Laser and ultrasound — Laser and ultrasound will be applied in group A as traditional method. On the other hand they will applied axillary in experimental groups
  Other Names: Post-isometric Facilitation

SUMMARY:
Elhafez Technique Combined with Dynamic Scapulohumeral Mobilization in Adhesive Capsulitis

DETAILED DESCRIPTION:
Elhafez Technique is an emerging rehabilitation approach that integrates axillary ultrasound, axillary laser therapy, and post-isometric facilitation (PIF) to target capsular stiffness, inflammation, and neuromuscular dysfunction. These techniques aim to enhance tissue healing, improve joint mobility, and reduce pain. When combined with Dynamic Scapulohumeral Mobilization (DSM), which focuses on restoring scapular control and shoulder joint biomechanics, this comprehensive approach may offer superior outcomes compared to conventional treatments.

This study aims to evaluate the biomechanical and functional effects of combining Elhafez Technique with DSM in patients with shoulder adhesive capsulitis. By assessing pain levels, ROM, and functional recovery, this research seeks to determine whether this combined intervention provides faster and more effective relief for patients suffering from this condition.

ELIGIBILITY:
Inclusion Criteria

1. Adults aged 30-60 years diagnosed with Stage 2 (Frozen) or Stage 3 (Thawing) Shoulder Adhesive Capsulitis based on American Shoulder and Elbow Surgeons (ASES) guidelines.
2. Pain score ≥4/10 on the Visual Analog Scale (VAS) for at least 3 months.
3. Restricted external rotation of ≥25% compared to the unaffected shoulder.
4. No prior shoulder injections, surgery, or physiotherapy within the last 3 months.

Exclusion Criteria

1. History of shoulder fractures, rotator cuff tears, or labral injuries.
2. Systemic inflammatory conditions (e.g., Rheumatoid Arthritis, Uncontrolled Diabetes).
3. Neurological disorders affecting the shoulder (e.g., Stroke, Parkinson's Disease).
4. Current participation in another physiotherapy intervent

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-09 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Range of motion | From enrollment to the end of treatment at 6 weeks
  Flexion, abduction and external rotation of the shoulder jooint

SECONDARY OUTCOMES:
Functional activities | From enrollment to the end of treatment at 6 weeks
  DASH will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Dokki, Giza, Giza Governorate, Egypt